CLINICAL TRIAL: NCT00450853
Title: Randomized Crossover Pharmacokinetic Evaluation of Subcutaneous Versus Intravenous Granisetron in Cancer Patients Treated With Platinum Based Chemotherapy
Brief Title: Randomized Crossover Pharmacokinetic Evaluation of Subcutaneous Versus Intravenous Granisetron in Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Principal Investigator, Jose Luis Perez Gracia, Main investigator, Clinica Universidad de Navarra, Universidad de Navarra
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GRA / SC-IV
Record Dates: First submitted 2007-03-21; First posted 2007-03-22 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Vomiting
Keywords: emesis; granisetron; pharmacokinetics; subcutaneous.
MeSH Terms: conditions — Vomiting | interventions — Granisetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Granisetron SC-Granisetron IV (Experimental): Granisetron SC followed by Granisetron IV
  Interventions: Drug: granisetron

INTERVENTIONS:
Drug: granisetron — Granisetron SC followed by granisetron IV
  Other Names: Granisetron SC followed by granisetron IV

SUMMARY:
Objective: to evaluate the bioavailability of subcutaneous granisetron.Patients receiving platinum-based chemotherapy will be randomized to receive granisetron 3 mg either subcutaneously or intravenously in a crossover manner during two cycles. Blood and urine samples will be collected after each cycle.

DETAILED DESCRIPTION:
5-HT3 antagonists are one of the mainstays of antiemetic treatment and they are administered either intravenously or orally. Nevertheless sometimes neither administration route is feasible, such as in patients unable to admit oral intake managed in an outpatient setting. Our objective is to evaluate the bioavailability of subcutaneous granisetron.Patients receiving platinum-based chemotherapy will be randomized to receive granisetron 3 mg either subcutaneously or intravenously in a crossover manner during two cycles. Blood and urine samples will be collected after each cycle. Pharmacokinetics of SC and IV granisetron will be prospectively compared.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients receiving platinum-based chemotherapy
* adequate bone marrow, hepatic and renal function, respectively defined by: platelets >100000/mm3 and absolute neutrophil count >1500/mm3; bilirubin, AST and ALT <2 times x upper limit of normality; and creatinine <1.5 mg/dl.
* ECOG performance status <2 and body mass index from 20-28 kg/m2.

Exclusion Criteria:

* Pregnancy
* Serious concomitant diseases, in the invesgator´s criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2005-04; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Bioavailability | Approximately 6 weeks

SECONDARY OUTCOMES:
Safety | Approximately 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso Gurpide, Principal Investigator — Oncology Department. Clinica Universitaria de Navarra
Locations (1):
- Clinica Universitaria de Navarra, Pamplona, Navarre, Spain